CLINICAL TRIAL: NCT01364246
Title: Phase I/II Study of Umbilical Cord Mesenchymal Stem Cell Therapy for Patients With Progressive Multiple Sclerosis and Neuromyelitis Optica
Brief Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Therapy for Patients With Progressive Multiple Sclerosis and Neuromyelitis Optica
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Beike Bio-Technology Co., Ltd. (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Nanjing Medical University (Other); Nanjing University Medical College Affiliated Wuxi Second Hospital (Unknown); Xuzhou Medical University (Other); The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BKCR-MS-1.0(2010)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Progressive Multiple Sclerosis; Neuromyelitis Optica.
Keywords: Progressive Multiple Sclerosis; neuromyelitis optica; Umbilical Cord Mesenchymal Stem Cell
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human umbilical cord mesenchymal stem cells transplantation (Experimental): Intervention group
  Interventions: Biological: human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells — Participants will be given hUC-MSCs transplantation.

SUMMARY:
Multiple sclerosis (MS) has been classically regarded as a chronic inflammatory autoimmune demyelinating disease of the central nervous system, along with a considerable pathological heterogeneity. Neuromyelitis optica (NMO) is a severe inflammatory, demyelinating disease, and its clinical characteristics include recurrent optic neuritis and longitudinally extensive transverse myelitis.

Current therapies provide only modest control of progressive Multiple Sclerosis and Neuromyelitis Optica.Stem cell therapy might open a light horizon in approaching to an efficient treatment in progressive MS and NMO. In this study, the safety and efficacy of Human Umbilical Cord Mesenchymal Stem Cells transplantation will be evaluated in patients with progressive MS and NMO.

ELIGIBILITY:
Inclusion Criteria:

* McDonald Diagnosis of Multiple Sclerosis or 2006 Diagnosis of neuromyelitis optica.
* Aged 16-65 years.
* Disease duration≥2years
* Poor response to steroid therapy.
* Written informed consent and follow the clinic trail procedure

Exclusion Criteria:

* Cardiac insufficiency; Renal insufficiency; hepatic insufficiency; Total bilirubin higher than 1.5 times of upper limit of normal value; AST /ALT higher than 2.5 times of upper limit of normal value.
* Combined Pneumonia or other Severe systemic bacteria infection.
* Severe drug allergic history or anaphylaxis to 2 or more food or medicine.
* Intracranial hypertension dues to Other brain lesions (eg. Brain cancer)/
* HIV+, TPPA +， patients diagnosed as HBV or HCV.
* Tumor Markers +
* Severe psychotic patients, cognitive dysfunction,Or can not understand or sign the Consent Form.
* Coagulation disorders.
* Uncontrolled hypertension after treatment，blood pressure≥180mmHg/110 mmHg.
* Pregnancy.
* Enrollment in other trials in the last 3 months.
* Other criteria the investigator consider improper for inclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-03 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Score of Expanded Disability Status Scale (EDSS) | 1 year after treatment

SECONDARY OUTCOMES:
Visual Evoked Potential (VEP) | 1 year after treatment
Brainstem Auditory Evoked Potential (BAEP) | 1 year after treatment
Somatosensory Evoked Potential(SEP) | 1 year after treatment
Brain Magnetic Resonance Imaging （MRI） Scan | 1 year after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing University Medical College Affiliated Drum Tower Hospital, Nanjing, Jiangsu, China